CLINICAL TRIAL: NCT00075387
Title: Phase II Clinical Trial of Patients With High-Grade Glioma Treated With Intra-Arterial Carboplatin-Based Chemotherapy, Randomized to Treatment With or Without Delayed Intravenous Sodium Thiosulfate as a Potential Chemoprotectant Against Severe Thrombocytopenia
Brief Title: Combination Chemotherapy With or Without Sodium Thiosulfate in Preventing Low Platelet Count While Treating Patients With Malignant Brain Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Edward Neuwelt, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00000922; NCI-2013-00781 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); eIRB #922 (Other: OHSU IRB); ONC-02019-L (Other: OHSU Knight Cancer Institute); CR00023930 (Other: OHSU IRB); MR00041590 (Other: OHSU IRB); CR00021317 (Other: OHSU IRB); CR00018679 (Other: OHSU IRB); CR00022743 (Other: OHSU IRB); IRB00000922 (Other: OHSU IRB)
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Malignant Glioma
MeSH Terms: conditions — Glioma | interventions — Carboplatin; Cyclophosphamide; etoposide phosphate; sodium thiosulfate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (combination chemotherapy) (Experimental): Patients receive cyclophosphamide IV, etoposide phosphate IV, and carboplatin IA over 10 minutes.
  Treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Cyclophosphamide; Drug: Etoposide Phosphate; Other: Quality-of-Life Assessment
- Arm II (combination chemotherapy, sodium thiosulfate) (Experimental): Patients receive cyclophosphamide IV, etoposide phosphate IV, and carboplatin IA as in Arm I. Patients also receive sodium thiosulfate IV over 15 minutes 4 and 8 hours later.
  Treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Cyclophosphamide; Drug: Etoposide Phosphate; Other: Quality-of-Life Assessment; Drug: Sodium Thiosulfate

INTERVENTIONS:
Drug: Carboplatin — Given IA
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Etoposide Phosphate — Given IV
  Other Names: Etopophos
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Sodium Thiosulfate — Given IV
  Other Names: Cyanide Antidote Package; Disodium Thiosulfate; S-Hydril; Sodium Hyposulfate; Sodium Thiosulfate Pentahydrate; Sodium Thiosulphate; Sodothiol; Thiosulfate, Sodium, Pentahydrate; Thiosulfuric acid disodium salt
  Arms: Arm II (combination chemotherapy, sodium thiosulfate)

SUMMARY:
This randomized phase II trial studies how well giving combination chemotherapy with or without sodium thiosulfate works in preventing low platelet count while treating patients with malignant brain tumors. Drugs used in chemotherapy, such as carboplatin, cyclophosphamide, and etoposide phosphate, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Sodium thiosulfate may prevent low platelet counts in patients receiving chemotherapy. It is not yet known whether combination chemotherapy is more effective with or without sodium thiosulfate in preventing low platelet count during treatment for brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the effect of delayed administration of sodium thiosulfate on the rates of platelet toxicity (i.e. platelet count less than 20,000), in subjects with high-grade glioma undergoing treatment with carboplatin, cyclophosphamide and etoposide/etoposide phosphate.

SECONDARY OBJECTIVES:

I. Assess tumor response in subjects with high-grade glioma undergoing treatment with carboplatin, cyclophosphamide and etoposide/etoposide phosphate, with or without delayed sodium thiosulfate.

II. Assess the effect of delayed administration of sodium thiosulfate on granulocyte and erythrocyte counts, in subjects undergoing treatment with carboplatin, cyclophosphamide and etoposide/etoposide phosphate.

III. Assess hearing changes, if any, at the higher frequencies in the standard testing range (4000 and 8000 Hertz [Hz]), and at higher frequencies above standard testing (9000 to 16000 Hz).

IV. Assess quality of life in subjects undergoing treatment with carboplatin, cyclophosphamide and etoposide phosphate.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive cyclophosphamide intravenously (IV), etoposide phosphate IV, and carboplatin intra-arterially (IA) over 10 minutes on day 1.

ARM II: Patients receive cyclophosphamide IV, etoposide phosphate IV, and carboplatin IA as in Arm I. Patients also receive sodium thiosulfate IV over 15 minutes 4 and 8 hours after carboplatin.

In both arms, treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically confirmed high-grade glioma are eligible; diagnosis of high-grade glioma will be made on the basis of needle biopsy, open biopsy, or surgical resection
* Subjects may have had prior focal or systemic radiation or chemotherapy; at least 14 days must have elapsed since radiation treatment and 28 days since prior chemotherapy
* Performance status (Eastern Cooperative Oncology Group [ECOG]) must be less than or equal to 2 (Karnofsky greater than or equal to 50)
* White blood cell count >= 2.5 x 10^3/mm^3
* Absolute granulocyte count >= 1.2 x 10^3/mm^3
* Platelets >= 100 x 10^3/mm^3
* Creatinine < 1.8
* Bilirubin < 2.0
* Baseline aspartate aminotransferase (AST)/alanine aminotransferase (ALT) serum glutamic oxaloacetic transaminase (SGOT)/serum glutamate pyruvate transaminase (SGPT) must be < 2.5 x institutional upper limits of normal
* Subject (or legal guardian) must sign a written informed consent in accordance with institutional guidelines
* Sexually active women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study treatment and for the duration of study treatment; should a female become pregnant or suspect she is pregnant while participating in this study, she should inform the investigator

Exclusion Criteria:

* Subjects with rapidly progressing central nervous system (CNS) disease with associated neurological deterioration
* Subjects with uncontrolled (over the last 30 days) clinically significant confounding medical conditions such as congestive heart failure
* Subjects who are pregnant, have a positive serum human chorionic gonadotropin (hCG) or are lactating
* Subjects who have contraindications to carboplatin, cyclophosphamide, etoposide phosphate, or sodium thiosulfate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2003-03-07 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of platelet toxicities (i.e. platelet count less than 20,000), graded according to the National Cancer Institute Common Toxicity Criteria version 3.0 | Up to 4 weeks after completion of study treatment
  The Pearson chi-square test will be the primary test to compare rates.

SECONDARY OUTCOMES:
Number of dose reductions and transfusions due to platelet toxicity | Up to 30 days after completion of study treatment
  Analyzed using generalized estimating equations and/or a generalized mixed model (for repeated measures analysis of variance) and the third using mixed model repeated measures analysis of variance model.
Tumor response (complete response + partial response + stable disease) assessed by neurologic exams, radiographic studies, and steroid dose | Up to 10 years
  The Pearson chi-square test will be the primary test to compare rates. Comparisons of rates will use the Pearson Chi-square test and logistic regression to adjust for potential confounders.
Time to response | Up to 10 years
  Descriptive summaries include Kaplan-Meier plots.
Time to disease progression | Up to 10 years
  Comparisons of time to disease progression will use the log rank test and the Cox proportional hazards model to adjust for potential confounders.
Granulocyte count | Up to 30 days after completion of study treatment
  The Pearson chi-square test will be the primary test to compare rates.
Erythrocyte counts | Up to 30 days after completion of study treatment
  The Pearson chi-square test will be the primary test to compare rates.
Change in hearing levels, if any, at the higher frequencies in the standard testing range (4000 and 8000 Hz), and at higher frequencies above standard testing (9000 to 16000 Hz) based on American Speech-Language-Hearing Association criteria | Baseline up to 30 days after completion of study treatment
  Descriptive summaries for hearing levels will include means by time and plots of hearing levels by patient over time. The analyses for hearing will include both a time to oto-toxicity (based on American Speech-Language-Hearing Association criteria) comparison using the log rank test and a repeated measure analysis of covariance of the actual hearing levels (with baseline hearing levels as the covariate). Separate analyses will be performed for each hearing frequency with no adjustment for multiple comparisons (as these analyses are descriptive in nature).
Quality of life assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 and Quality of Life Questionnaire-Brain Module-20 | Up to 60 days after completion of study treatment
  Summarized by means over time and by plots of values over time for each patient. Quality of life data comparisons between the groups will use repeated measure analysis of covariance (baseline assessment as the covariate).

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Neuwelt, Principal Investigator — OHSU Knight Cancer Institute
Locations (3):
- United States (3):
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - OHSU Knight Cancer Institute, Portland, Oregon